CLINICAL TRIAL: NCT00698425
Title: Single Center, Single-masked, Randomized, Dose Escalation Study to Evaluate Safety and Tolerability of Transscleral Iontophoresis Using Citrate Buffer Delivered by the EyeGate® II Drug Delivery Device System in Healthy Adult Volunteers
Brief Title: Safety and Tolerability Study of Transscleral Iontophoresis by the EyeGate® II Drug Delivery Device System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Stephen From, President and Chief Executive Officer, Eyegate Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/Eyegate/01
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Iontophoresis; Ophthalmology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (19):
- 1: 0 mA-min (0 mA for 4 min) (Experimental): Ocular iontophoresis 0 mA-min (0 mA for 4 minutes)
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 2: 4 mA-min (2 mA for 2 min), + polarity (Experimental): Ocular iontophoresis 4 mA-min (2 mA for 2 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 3: 5 mA-min (2.5 mA for 2 min), + (Experimental): Ocular iontophoresis 5 mA-min (2.5 mA for 2 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 4: 6 mA-min (3 mA for 2 min), + polarity (Experimental): Ocular iontophoresis 6 mA-min (3 mA for 2 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 5: 7 mA-min (3.5 mA for 2 min), + (Experimental): Ocular iontophoresis 7 mA-min (3.5 mA for 2 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 6: 8 mA-min (4 mA for 2 min), + polarity (Experimental): Ocular iontophoresis 8 mA-min (4 mA for 2 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 7: 7 mA-min (3.5 mA for 2 min), - (Experimental): 7 mA-min (3.5 mA for 2 minutes), negative polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 8: 8 mA-min (4 mA for 2 min), - polarity (Experimental): Ocular iontophoresis 8 mA-min (4 mA for 2 minutes), negative polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 9: 20 mA-min (4 mA for 5 min), + (Experimental): Ocular iontophoresis 20 mA-min (4 mA for 5 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 10: 20 mA-min (2 mA for 10 min), + (Experimental): Ocular iontophoresis 20 mA-min (2 mA for 10 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 11: 20 mA-min (4 mA for 5 min), - (Experimental): Ocular iontophoresis 20 mA-min (4 mA for 5 minutes), negative polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 12: 20 mA-min (2 mA for 10 min), - (Experimental): Ocular iontophoresis 20 mA-min (2 mA for 10 minutes), negative polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 13: 0 mA-min (0 mA for 10.5 min) (Experimental): Ocular iontophoresis 0 mA-min (0 mA for 10.5 minutes)
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 14: 13.5 mA-min (4.5 mA for 3 min), + (Experimental): Ocular iontophoresis 13.5 mA-min (4.5 mA for 3 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 15: 15 mA-min (5 mA for 3 min), + (Experimental): Ocular iontophoresis 15 mA-min (5 mA for 3 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 16: 16.5 mA-min (5.5 mA for 3 min), + (Experimental): Ocular iontophoresis 16.5 mA-min (5.5 mA for 3 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 17: 18 mA-min (6 mA for 3 min), + (Experimental): Ocular iontophoresis 18 mA-min (6 mA for 3 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 18: 19.5 mA-min (6.5 mA for 3 min), + (Experimental): Ocular iontophoresis 19.5 mA-min (6.5 mA for 3 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer
- 19: 20 mA-min (7 mA for 3.84 min), + (Experimental): Ocular iontophoresis 20 mA-min (7 mA for 3.84 minutes), positive polarity
  Interventions: Other: EyeGate II® Drug Delivery System; Drug: Citrate buffer

INTERVENTIONS:
Other: EyeGate II® Drug Delivery System — Transscleral iontophoresis using citrate buffer delivered by EyeGate II® Drug Delivery System
  Other Names: Citrate buffer
Drug: Citrate buffer — Transscleral iontophoresis using citrate buffer delivered by EyeGate II® Drug Delivery System

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single iontophoretic dose of buffered solution administered through the EyeGate® II Drug Delivery System in healthy adult human volunteers.

DETAILED DESCRIPTION:
This is a single center, randomized, single-masked, comparative group, safety and tolerability study of single dose levels of citrate buffer delivered through transcleral iontophoresis administered via the EyeGate® II Drug Delivery System. The current study will also determine the safety and tolerability of the dose ranges of transcleral iontophoresis from 2 mA through 7 mA and will determine the safety and tolerability of the application of the Eyegate II system on the eye for time ranges of up to 10.5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Normal ophthalmic examination in both eyes

Exclusion Criteria:

* Presence of subjective ocular symptoms
* Presence of conjunctival hyperemia, chemosis, watering, conjunctival discharge
* Ocular trauma

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety assessed through patient reported adverse events | Prospective

SECONDARY OUTCOMES:
Ophthalmic examinations | Prospective
Ocular discomfort on a visual analog scale (VAS) | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Manjoo Reddy, MS, Principal Investigator — St Johns Medical College Hospital, Bangalore, India
Locations (1):
- St. John's Medical College Hospital, Bangalore, Karnataka, India